CLINICAL TRIAL: NCT07308015
Title: Clinical Study on the Treatment of Rhinitis Sicca With Sodium Hyaluronate Adjustable Nasal Irrigator
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: China-Japan Union Hospital (Other)
Responsible Party: Principal Investigator, Dongdong Zhu, China-Japan Union Hospital, China-Japan Union Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025052906
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Rhinitis Sicca

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Physiological seawater adjustable nasal irrigator
  Interventions: Drug: Physiological seawater adjustable nasal irrigator
- Experimental group (Experimental): Sodium hyaluronate adjustable nasal irrigator
  Interventions: Drug: Sodium hyaluronate adjustable nasal irrigator

INTERVENTIONS:
Drug: Physiological seawater adjustable nasal irrigator — Nasal spray of Physiological seawater.
  Arms: Control group
Drug: Sodium hyaluronate adjustable nasal irrigator — Nasal spray of Sodium hyaluronate
  Arms: Experimental group

SUMMARY:
To observe the therapeutic effect of sodium hyaluronate adjustable nasal irrigator on various types of rhinitis sicca and compare it with the therapeutic effect of the commonly used physiological seawater nasal spray in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms: Dry nose sensation, little and thick nasal discharge, nosebleeds, itchy nasal cavity, and dryness in the nasopharynx. Physical signs: Nasal endoscopy often reveals dry and congested nasal mucosa, which appears grayish-white or dark red, losing its normal luster. There are often dry, thick secretions, scabs or blood scabs on it. The surface of the nasal mucosa is eroded and ulcers occur. The mucosal lesions are most obvious in the anterior part of the nasal cavity. A diagnosis can be made if one or more of the above symptoms and signs are present.

Exclusion Criteria:

1. Those with dry rhinitis and chronic inflammation of the lower respiratory tract.
2. Those confirmed by examination to be caused by certain latent lesions in the mouth, nose, throat, esophagu.s, neck or the whole body
3. Those who have used drugs for treating dry rhinitis or other medications within the past 30 days.
4. Pregnant or lactating women.
5. Those who are allergic to this medicine.
6. Those with severe cardiovascular, liver, kidney and hematopoietic system diseases, etc.
7. Mentally ill patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-06-12 (Estimated); Study Completion 2026-06-12 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Two weeks after the treatment

SECONDARY OUTCOMES:
Nasal endoscopy examination score | Two weeks after the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Union Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Undecided